CLINICAL TRIAL: NCT05849103
Title: Comprehensive Postpartum Management for Women With Hypertensive Disorders of Pregnancy: A Randomized Controlled
Brief Title: Comprehensive Postpartum Management for Women With Hypertensive Disorders of Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Sarah Osmundson, MD, MS (Unknown); Alex Phelps, MD (Unknown); Julia Phillippi, PhD, CNM (Unknown); Soha Patel, MD, MSPH (Unknown); Etoi Garrison, MD, PhD (Unknown); Kathryn Lindley, MD (Unknown)
Responsible Party: Principal Investigator, Sarah Osmundson, Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: R21NR020857-01 (NIH)
Record Dates: First submitted 2023-04-10; First posted 2023-05-08 (Actual); Results first posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Hypertension, Pregnancy-Induced; Postpartum Preeclampsia; Hypertension; Maternal
Keywords: Hypertension; Postpartum hypertension
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Hypertension

STUDY DESIGN:
Intervention Model Description: A factorial study design will be used where participants will be randomized in a 1:1:1:1 ratio to two intervention types (blood pressure target, hypertension care model) or four total interventions.
Who Masked: Outcomes Assessor
Masking Description: Research personnel assessing outcomes will be masked to the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A) Standard BP Control, Clinician Monitoring (Active Comparator): Target blood pressure will be less than 150/100. Participants will be instructed to check their blood pressures twice a day for two weeks and daily for weeks 3-6 after delivery and report abnormal blood pressures or symptoms to their obstetric clinicians. Additional postpartum visits beyond the blood pressure check will be directed by their obstetric clinician.
  Interventions: Other: Blood Pressure Control Targets; Other: Hypertension Management
- B) Tight BP Control, Clinician Monitoring (Active Comparator): Target blood pressure will be less than 140/90. Participants will be instructed to check their blood pressures twice a day for two weeks and daily for weeks 3-6 after delivery and report abnormal blood pressures or symptoms to their obstetric clinicians. Additional postpartum visits beyond the blood pressure check will be directed by their obstetric clinician.
  Interventions: Other: Blood Pressure Control Targets; Other: Hypertension Management
- C) Standard BP Control, Care Navigation (Active Comparator): Target blood pressure will be less than 150/100. Participants will check blood pressures twice daily for 14 days and daily for weeks 3-6. A nurse navigator will review their blood pressures M-F for Weeks 1-2 and weekly for weeks 3-6 and will provide feedback on blood pressure values and recommend initiating or escalating medications as needed. The nurse navigator will communicate progress to the participant's clinicians and will remind the participant of their appointments. The nurse navigator will facilitate a visit around 3 months with a primary care clinician or a cardiologist for hypertension follow up.
  Interventions: Other: Blood Pressure Control Targets; Other: Hypertension Management
- D) Tight BP Control, Care Navigation (Active Comparator): Target blood pressure will be less than 140/90. Participants will check blood pressures twice daily for 14 days and daily for weeks 3-6. A nurse navigator will review their blood pressures M-F for Weeks 1-2 and weekly for weeks 3-6 and will provide feedback on blood pressure values and recommend initiating or escalating medications as needed. The nurse navigator will communicate progress to the participant's clinicians and will remind the participant of their appointments. The nurse navigator will facilitate a visit around 3 months with a primary care clinician or a cardiologist for hypertension follow up.
  Interventions: Other: Blood Pressure Control Targets; Other: Hypertension Management

INTERVENTIONS:
Other: Blood Pressure Control Targets — This intervention specifies the goal blood pressure as less than 150/100 versus less than 140/90
Other: Hypertension Management — This intervention specifies whether the participant has hypertension management through their obstetric clinician or through a single nurse navigator who provides feedback and modifies hypertension treatment based on blood pressure values submitted by the participant.

SUMMARY:
Investigators propose a comprehensive management program for postpartum patients with HDP who are at risk for severe maternal morbidity and mortality. Our program will emphasize three key components: 1) self-monitoring of blood pressures with app-based reporting connected to our electronic health record, 2) blood pressure management directed by a program navigator with guideline and physician support and 3) facilitated transitions of care to primary care clinicians for hypertension management. Investigators will randomize 300 patents with HDP on postpartum day one with follow up through 3 months postpartum. Primary outcome will be blood pressure reporting at 7-10 postpartum. Secondary outcomes include blood pressure control at 7-10 days postpartum, identification and treatment of severe blood pressures, severe maternal morbidity, hospital readmission, triage visits for hypertension, postpartum and primary care visit attendance, and multiple patient-reported outcome measures. All outcomes will be stratified by race (Black and non-Black) to evaluate disparities and by tight versus usual blood pressure control to evaluate the impact of strict postpartum blood pressure control on outcomes. Investigators hypothesize that a comprehensive postpartum HDP management program will improve hypertension control for all patients and reduce disparities that affect Black patients, and that stricter blood pressure control will be associated with fewer adverse outcomes.

DETAILED DESCRIPTION:
Hypertension complicates 10% of pregnancies in the U.S., directly accounting for 7% of pregnancy-related deaths and 38% of severe maternal morbidity. Hypertensive disorders of pregnancy (HDP) include chronic hypertension, gestational hypertension, preeclampsia, hemolysis-elevated-liver enzymes-low platelets (HELLP), and eclampsia, and occur 2.5 times more frequently among Black compared to non-Black patients. The weeks after delivery are crucial for maternal health, severe maternal morbidity, and hypertension-associated morbidity. Half of all pregnancy-related deaths occur in this time and Black patients are impacted disproportionally by these morbidities including pulmonary edema, stroke, and renal failure.

The American College of Obstetricians and Gynecologists (ACOG) recently redefined postpartum care to encompass 12 months after birth and stressed the importance of connecting postpartum patients to primary care clinicians to manage chronic conditions. This handoff is critical as 50% of patients with HDP develop chronic hypertension, and patients affected by HDP have twice the risk of later cardiovascular-related death. Recently, Tennessee expanded Medicaid coverage to 12 months postpartum. Given that most obstetric clinicians do not provide comprehensive primary care, investigators urgently need models for bridging gaps in care after pregnancy. While interventions such as telemedicine and peer navigation demonstrate promise to improve patient engagement in care and reduce postpartum racial disparities,15-18 no randomized trials address system-level initiatives to improve postpartum care for patients with HDP.

Another area of active investigation relates to establishing appropriate blood pressure targets for patients in and around the time of pregnancy. Recent findings from the Chronic Hypertension and Pregnancy Trial suggest that stricter control of antepartum blood pressure is beneficial in reducing the incidence of a composite adverse perinatal outcome which included preeclampsia with severe features, medically indicated preterm birth at less than 35 weeks of gestation, placental abruption, and fetal or neonatal death. This trial has been practice-changing, lowering the historic antepartum blood pressure target from 160/110mmHg (millimeter of mercury) to less than 140/90mmHg. However, this trial did not contemplate the management of maternal blood pressure in the postpartum period. ACOG presently endorses a postpartum goal of less than 150/100mmHg which, notably, is higher than the newly established antepartum goal. Furthermore, the blood pressure target set for non-pregnant adults by the American College of Cardiology and American Heart Association is even lower, at less than 120/80mmHg to minimize the cardiovascular disease risk associated with chronic hypertension.

Investigators propose a comprehensive management program for postpartum patients with HDP who are at risk for severe maternal morbidity and mortality. Our program will emphasize three key components: 1) self-monitoring of blood pressures with app-based reporting connected to our electronic health record, 2) blood pressure management directed by a program navigator with guideline and physician support and 3) facilitated transitions of care to primary care clinicians for hypertension management. Investigators will randomize 300 patents with HDP on postpartum day one with follow up through 3 months postpartum. Primary outcome will be blood pressure reporting at 7-10 postpartum. Secondary outcomes include blood pressure control at 7-10 days postpartum, identification and treatment of severe blood pressures, severe maternal morbidity, hospital readmission, triage visits for hypertension, postpartum and primary care visit attendance, and multiple patient-reported outcome measures. All outcomes will be stratified by race (Black and non-Black) to evaluate disparities and by tight versus usual blood pressure control to evaluate the impact of strict postpartum blood pressure control on outcomes. Investigators hypothesize that a comprehensive postpartum HDP management program will improve hypertension control for all patients and reduce disparities that affect Black patients, and that stricter blood pressure control will be associated with fewer adverse outcomes.

ELIGIBILITY:
Inclusion Criteria

1. Age >18 years
2. Diagnosed with a Hypertensive Disorder of Pregnancy (HDP), which includes chronic hypertension, preeclampsia, gestational hypertension, HELLP Syndrome (Hemolysis, Elevated Liver enzymes, Low Platelets), or eclampsia (O10, O11, O13, O14, O15, O16) Exclusion Criteria

1. Not able or willing to receive electronic surveys 2. Deemed inappropriate for study enrollment by the bedside nurse 3. Non-English speaking 4. Contraindication to ACOG-recommended hypertension control (i.e. chronic kidney disease, stroke)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who have recently given birth. The aim of this study evaluate post-partum hypertension care.
Enrollment: 343 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Osmundson, MD, Principal Investigator — Associate Professor Maternal-Fetal Medicine
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | A) Standard BP Control, Clinician Monitoring | B) Tight BP Control, Clinician Monitoring | C) Standard BP Control, Care Navigation | D) Tight BP Control, Care Navigation
Started | 86 | 86 | 86 | 85
Completed | 84 | 83 | 82 | 85
Not Completed | 2 | 3 | 4 | 0

BASELINE CHARACTERISTICS:
Population: Median (Interquartile Range)
Groups:
- Total: Total of all reporting groups
Arm/Group | A) Standard BP Control, Clinician Monitoring | B) Tight BP Control, Clinician Monitoring | C) Standard BP Control, Care Navigation | D) Tight BP Control, Care Navigation | Total
Number analyzed (Participants) | 84 | 82 | 83 | 85 | 334
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Continuous age in years
  years | 29.0 [22.0 to 33.5] | 30.5 [27.0 to 34.0] | 30.0 [24.0 to 35.0] | 30.0 [26.0 to 34.0] | 30.0 [25.0 to 34.0]
Sex: Female, Male [Count of Participants; unit: Participants] — Percentage male and female
  Participants
    Female | 84 | 82 | 83 | 85 | 334
    Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race or Ethnicity: Asian | 2 | 4 | 0 | 2 | 8
  Race or Ethnicity: Hispanic | 11 | 0 | 8 | 7 | 26
  Race or Ethnicity: Multi-racial | 5 | 4 | 2 | 5 | 16
  Race or Ethnicity: Non-Hispanic Black | 21 | 20 | 24 | 24 | 89
  Race or Ethnicity: Non-Hispanic White | 43 | 49 | 47 | 45 | 184
  Race or Ethnicity: Unknown | 2 | 5 | 2 | 2 | 11
Region of Enrollment [Number; unit: participants]
  United States | 84 | 82 | 83 | 85 | 334

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Recorded Blood Pressure Values in Office
Description: Proportion of participants with blood pressure values recorded in the office
Time Frame: 7-10 days post delivery
Measure: Count of Participants; unit: Participants
Arm/Group | A) Standard BP Control, Clinician Monitoring | B) Tight BP Control, Clinician Monitoring | C) Standard BP Control, Care Navigation | D) Tight BP Control, Care Navigation
Number analyzed (Participants) | 84 | 82 | 83 | 85
Participants | 43 | 44 | 49 | 56

2. Secondary Outcome: Proportion of Participants With Recorded Blood Pressure Values, Any Reporting
Description: Proportion of participants with blood pressure values recorded through any means
Time Frame: 7-10 days post delivery
Measure: Number; unit: participants
Arm/Group | A) Standard BP Control, Clinician Monitoring | B) Tight BP Control, Clinician Monitoring | C) Standard BP Control, Care Navigation | D) Tight BP Control, Care Navigation
Number analyzed (Participants) | 84 | 82 | 83 | 85
participants | 48 | 47 | 76 | 78

3. Secondary Outcome: Systolic Blood Pressure, 7-10 Days
Description: Mean difference in systolic blood pressure from baseline, 7-10 days
Time Frame: 7-10 days post delivery
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | A) Standard BP Control, Clinician Monitoring | B) Tight BP Control, Clinician Monitoring | C) Standard BP Control, Care Navigation | D) Tight BP Control, Care Navigation
Number analyzed (Participants) | 84 | 82 | 83 | 85
mmHg | 130 [122 to 139] | 132 [125 to 138] | 128 [123 to 136] | 128 [120 to 137]

4. Secondary Outcome: Diastolic Blood Pressure
Description: Mean difference in diastolic blood pressure from baseline, 7-10 days
Time Frame: 7-10 days post delivery
Population: Participants
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | A) Standard BP Control, Clinician Monitoring | B) Tight BP Control, Clinician Monitoring | C) Standard BP Control, Care Navigation | D) Tight BP Control, Care Navigation
Number analyzed (Participants) | 84 | 82 | 83 | 85
mmHg | 84 [78 to 90] | 82 [78 to 90] | 84 [78 to 89] | 84 [78 to 90]

5. Secondary Outcome: Systolic Blood Pressure, 4-6 Weeks
Description: Mean difference in systolic blood pressure from baseline, 4-6 weeks
Time Frame: 4-6 weeks post delivery
Reporting Status: Not Posted, anticipated posting 2026-01

6. Secondary Outcome: Diastolic Blood Pressure, 4-6 Weeks
Description: Mean difference in diastolic blood pressure from baseline, 4-6 weeks after delivery
Time Frame: 4-6 weeks post delivery
Reporting Status: Not Posted, anticipated posting 2026-01

7. Secondary Outcome: Initiated New Medications
Description: Initiated new antihypertensive medications by 7-10 days postpartum
Time Frame: 7-10 days
Population: Participants
Measure: Count of Participants; unit: Participants
Arm/Group | A) Standard BP Control, Clinician Monitoring | B) Tight BP Control, Clinician Monitoring | C) Standard BP Control, Care Navigation | D) Tight BP Control, Care Navigation
Number analyzed (Participants) | 41 | 45 | 49 | 53
Participants | 9 | 7 | 4 | 17

8. Secondary Outcome: Sustained Severe Hypertension, 7-10 Days
Description: Proportion of participants with two blood pressures >=160/100 at least 15 minutes apart
Time Frame: 7-10 days postpartum
Population: Participants
Measure: Count of Participants; unit: Participants
Arm/Group | A) Standard BP Control, Clinician Monitoring | B) Tight BP Control, Clinician Monitoring | C) Standard BP Control, Care Navigation | D) Tight BP Control, Care Navigation
Number analyzed (Participants) | 80 | 75 | 80 | 81
Participants | 6 | 5 | 6 | 9

9. Secondary Outcome: Unplanned Visits
Description: Proportion of patients with obstetric triage visits, emergency department visits, or hospital readmission
Time Frame: 7-10 days
Population: Participants
Measure: Count of Participants; unit: Participants
Arm/Group | A) Standard BP Control, Clinician Monitoring | B) Tight BP Control, Clinician Monitoring | C) Standard BP Control, Care Navigation | D) Tight BP Control, Care Navigation
Number analyzed (Participants) | 84 | 82 | 83 | 85
Participants | 13 | 10 | 10 | 12

10. Secondary Outcome: Postpartum Visit Attendance
Description: Proportion of patients with postpartum visit attendance
Time Frame: 3-6 weeks post delivery
Reporting Status: Not Posted, anticipated posting 2026-01

11. Secondary Outcome: Primary Care Visit Attendance
Description: Proportion of patients with primary care visit attendance
Time Frame: 3 months post delivery
Reporting Status: Not Posted, anticipated posting 2026-01

12. Other Pre Specified Outcome: Feeling That Their Voice is Heard
Description: Proportion of patients who respond 'yes' to feeling that their voice is heard
Time Frame: 2 weeks post delivery
Reporting Status: Not Posted, anticipated posting 2026-01

13. Other Pre Specified Outcome: Perceived Stress
Description: mean T-score (Range 1-100) using NIH Toolbox
Time Frame: 2 weeks post delivery
Reporting Status: Not Posted, anticipated posting 2026-01

14. Other Pre Specified Outcome: Self-Efficacy
Description: mean T-score (Range 1-100) on Self-efficacy PROMIS measure
Time Frame: 2 weeks post delivery
Reporting Status: Not Posted, anticipated posting 2026-01

15. Other Pre Specified Outcome: Mothers on Respect Index Score
Description: mean score (range 14-84) for the Mothers on Respect Index Score
Time Frame: 6 weeks post delivery
Reporting Status: Not Posted, anticipated posting 2026-01

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 year.
Arm/Group | A) Standard BP Control, Clinician Monitoring | B) Tight BP Control, Clinician Monitoring | C) Standard BP Control, Care Navigation | D) Tight BP Control, Care Navigation
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/82 | 0/83 | 0/85
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/82 | 0/83 | 0/85
Other Adverse Events (participants affected / at risk) | 0/84 | 0/82 | 0/83 | 0/85

LIMITATIONS AND CAVEATS:
There are important limitations to our study. First, the randomized controlled trial design increases internal validity of our findings but can also decrease external validity. Forty-eight percent of eligible patients did not enroll, raising concerns for how our interventions would perform outside of a research setting. In addition, we were unable to enroll non-English speaking participants, who are an important population to consider especially for larger implementation efforts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/03/NCT05849103/Prot_SAP_ICF_000.pdf